CLINICAL TRIAL: NCT04989075
Title: Effect of Oral Prophylactic Measures on the Occurrence of Pre-eclampsia (OP-PE) in High-risk Pregnant Women: A Cluster-randomized Controlled Trial
Brief Title: Oral Prophylactic Measures on the Occurrence of Pre-eclampsia (OP-PE)
Acronym: OP-PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Collaborators: Cheikh Anta Diop University, Senegal (Other); University of Ouagadougou, Burkina Faso (Other)
Responsible Party: Principal Investigator, Carrouel Florence, Associate professor, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OP-PE
Record Dates: First submitted 2021-07-19; First posted 2021-08-04 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Complications
Keywords: pre-eclampsia; pregnant; periodontal disease; interdental microbiota
MeSH Terms: conditions — Pregnancy Complications; Pre-Eclampsia; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: This trial is designed as an two-arm parallel cluster randomized controlled trial with antenatal obstetric clinic as the unit of randomisation and an allocation ratio of 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will continue its usual oral hygiene practice.
- Oral prophylactic intervention (Experimental): For the study group, the oral prophylactic intervention will consist of provision of specfic package including soft-bristled manual toothbrush, toothpaste, and a kit of calibrated interdental brushes (IDBs)(Curaprox CPS; Curaden) of sizes corresponding to the diameter of their interdental spaces. The participants will be instructed to brush their teeeth twice-daily and to realise a daily interdental brushing until delivery. The instructions for the use of the toothbrush and IDBs comprised verbal instructions supported by practical demonstration. The first use of the material will be conducted under the supervision of a qualified public health professor.
  Interventions: Other: Oral prophylactic intervention

INTERVENTIONS:
Other: Oral prophylactic intervention — The oral prophylactic intervention will consist of the provision of specific package including a soft-bristled manual toothbrush, toothpaste, and a kit of calibrated interdental brushes (IDBs)(Curaprox CPS; Curaden) of sizes corresponding to the diameter of their interdental spaces. The participants will be instructed to brush their teeeth twice-daily and to realise a daily interdental brushing until delivery. The instructions for the use of the toothbrush and IDBs comprised verbal instructions supported by practical demonstration. The first use of the material will be conducted under the supervision of a qualified public health professor.
  Arms: Oral prophylactic intervention

SUMMARY:
Pre-eclampsia (PE) remains a major source of maternal and perinatal morbidity and mortality especially in low- and middle-income settings. PE, a pregnancy-specific hypertensive disorder, characterized by the development of placental endothelial dysfunction resulting in, among the most common diagnostic features, concomitant hypertension and proteinuria that may evolve into organs with fluctuating clinical specificities. Current studies indicate that periodontal disorders during pregnancy and particularly periodontal pathogens may be related to the risk of PE. Standard oral hygiene methods, based mainly on the joint use of toothbrushes and interdental brushes, reduce periodontal inflammatory risk, modulate of the dysbiotic oral microbiome. The purpose of the present study is to compare the PE outcomes in high-risk pregnant women receiving oral prophylactic measures to a control group. One specific question is addressed as follows according to the PICO principles: In high-risk pregnant women (Population), does oral prophylactic measures (Intervention) have a beneficial effect on PE parameters (Outcome) compared to pregnant women without any specific oral prophylactic measures (Control)?

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman
* women from sub-Saharan Africa
* aged from 18 to 40 years old
* nullipares at the time of the obstetrical consultation
* up to 12 weeks pregnant
* acceptance of the terms and conditions of the study
* signature of the informed consent form,

Exclusion Criteria:

* fetal distress
* congenital uterine and vaginal abnormalities
* infectious or systemic diseases such as HIV, tuberculosis, candidiasis, cancers, hemopathies
* premature termination of pregnancy for medical reasons
* diagnosis of periodontitis defined as interproximal CAL ≥1 mm at ≥2 non-adjacent teeth, or buccal/oral CAL ≥3 mm with probing depth >3 mm at ≥2 teeth, not attributable to non-periodontitis-related causes
* history or treatment of PD
* a course of dental or orthodontic treatment
* absence of the 4 premolar-molar pairs
* less than 20 natural teeth, excluding third molars
* medication affecting the gum and/or oral mucosa
* regularly using interdental brushes and/or dental floss and/or mouthwash
* unable to answer questions or non-cooperative.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of pre-eclampsia from baseline during the pregnancy | 9 months of pregnancy
  To determine if pregnant women suffer from pre-eclampsia, several indices are measured (diastolic or systolic pressure and proteinuria or urinary protein/creatinine ratio).
  The combination of the results of pressure and proteinuria permits to classify of a woman as suffering from pre-eclampsia if:
  1. the diastolic pressure is higher than 90 mm Hg on two 4 hours intervals, or > 110 mm Hg once, or systolic pressure > 140 mm Hg on two 4 hours intervals, or > 160 mm Hg once, after 20 weeks of gestation and,
  2. the proteinuria measured is of 2+ or more, or > 300mg/24 hours, or > 500mg/L or urinary protein/creatinine ratio > 0.034g/mmol.

SECONDARY OUTCOMES:
Number of pathogenic bacteria in the interdental microbiota during the pregnancy | 3, 4, 6 and 8 months of pregnancy
  Quantitative PCR experiments will be performed and a quantitative analysis of the interdental microbiota will be made
Change of bleeding on probing during the pregnancy | 3, 4, 6 and 8 months of pregnancy
  Quantification of the bleeding on probing of the teeth with a periodontal probe
Change of pocket probing depth of teeth during the pregnancy | 3, 4, 6 and 8 months of pregnancy
  Quantification of the pocket probing depth of the teeth with a periodontal probe
Change of clinical attachment level of teeth during the pregnancy | 3, 4, 6 and 8 months of pregnancy
  Quantification of the clinical attachment level of the teeth with a periodontal probe
Change of gingival index of teeth during the pregnancy | 3, 4, 6 and 8 months of pregnancy
  Quantification of the gingival index

CONTACTS AND LOCATIONS:
Overall Officials: Florence Carrouel, Dr, Study Director — P2S, UR4129, University of Lyon
Locations (1):
- Hospital, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gare J, Kanoute A, Meda N, Viennot S, Bourgeois D, Carrouel F. Periodontal Conditions and Pathogens Associated with Pre-Eclampsia: A Scoping Review. Int J Environ Res Public Health. 2021 Jul 5;18(13):7194. doi: 10.3390/ijerph18137194. PMID 34281133
- [Derived] Carrouel F, Kanoute A, Faye D, Mazur M, Perrier H, Vitiello F, Ardan R, Clement C, Lan R, Bourgeois D. Impact of Interdental Brushing on Pregnancy-Associated Gingivitis: A Secondary Analysis of a Randomised Controlled Trial. J Clin Periodontol. 2026 Jan 20. doi: 10.1111/jcpe.70085. Online ahead of print. PMID 41558746